CLINICAL TRIAL: NCT00492895
Title: Photosensitivity of the Skin Under Azathioprin in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007DR2040
Record Dates: First submitted 2007-06-19; First posted 2007-06-27 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): one arm only. Crossover study
  Interventions: Drug: Discontinuation of Azathioprin

INTERVENTIONS:
Drug: Discontinuation of Azathioprin — Discontinuation of Azathioprin

SUMMARY:
Photosensitivity of the skin to UVA and UVB will be determined

DETAILED DESCRIPTION:
Photosensitivity of the skin to UVA and UVB in renal transplant recipients with and without azathioprine will be determined. Azathioprine will be discontinued and photosensitivity determined after a wash-out period of three months

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Renal transplant recipients under azathioprin

Exclusion criteria:

* Treatment with Prograf (Tacrolimus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Photosensitivity of the skin to UVA and UVB | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, M.D, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- Clinic for Dermatology, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Result] Hofbauer GF, Attard NR, Harwood CA, McGregor JM, Dziunycz P, Iotzova-Weiss G, Straub G, Meyer R, Kamenisch Y, Berneburg M, French LE, Wuthrich RP, Karran P, Serra AL. Reversal of UVA skin photosensitivity and DNA damage in kidney transplant recipients by replacing azathioprine. Am J Transplant. 2012 Jan;12(1):218-25. doi: 10.1111/j.1600-6143.2011.03751.x. Epub 2011 Sep 22. PMID 21943390